CLINICAL TRIAL: NCT00000294
Title: Effects of Carvedilol on Cocaine Use in Humans
Brief Title: Effects of Carvedilol on Cocaine Use in Humans - 11
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Minnesota (Other)
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09259-11; P50-09259-11
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1999-03

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Carvedilol

INTERVENTIONS:
Drug: Carvedilol

SUMMARY:
The purpose of this study is to examine carvedilol effects in response to cocaine.

DETAILED DESCRIPTION:
The purpose of this study was to determine whether carvedilol, and alpha and beta adrenergic blocker, would inhibit the priming effect of cocaine in a laboratory model. A total of 12 subjects were enrolled in this double blind, placebo controlled, outpatient study. After an adaptation session, three experimental sessions were held, 2-9 days apart. On each of 3 experimental sessions, a single oral dose of low (25mg) or high dose of carvedilol (50mg) or placebo were administered. Two hours following carvedilol or placebo treatment, subjects received a priming dose of smoked cocaine, 0.4 mg/kg. during the second part of the session, subjects had the option to earn up to 2 tokens by working on a computer task that could later be exchanged for money or deliveries of cocaine. We proposed that blockage of adrenergic receptors by carvedilol would significantly alter the subjective and physiological effects of cocaine.

ELIGIBILITY:
Inclusion Criteria:

Male/Female between 20 and 55. History of smoked or intravenous cocaine use on the average of at least once a week over a 6 month period. current history of good health and normal EKG. Not pregnant as determined by pregnancy screening nor breast feeding, using acceptable birth control methods (e.g. birth control pills diaphragm, condoms plus foam)

Exclusion Criteria:

Current problems with major psychiatric illnesses including bipolar disorder, schizophrenia, or anxiety disorders. History of major medical illnesses including asthma and chronic obstructive pulmonary disease. Currently on a drug related parole or probation. Treated for chemical dependency withing the past 6 months.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1998-09; Study Completion 2001-12

PRIMARY OUTCOMES:
Behavioral
Subjective
Physiologic measures

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States